CLINICAL TRIAL: NCT01511003
Title: An Open- Label, Single-arm, Phase 4 Study to Assess the Efficacy and Safety of Tacrolimus in Active Rheumatoid Arthritis Patients Shown Unsuccessful Response Against DMARDs
Brief Title: A Study is to Assess Efficacy and Safety of Tacrolimus in Active Rheumatoid Arthritis Patients Who Showed Unsuccessful Response to Existing Disease Modifying Antirheumatic Drugs (DMARDs)
Acronym: TREASURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRGRA-10-04-KOR
Record Dates: First submitted 2012-01-04; First posted 2012-01-18 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: calcineurin inhibitor; Prograf; Rheumatoid arthritis (RA); Tacrolimus
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus group (Experimental): oral
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf

SUMMARY:
This study is to assess efficacy and safety of tacrolimus in active rheumatoid arthritis patients who showed unsuccessful response to existing DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have rheumatoid arthritis for 6 months or longer based on American College of Rheumatology (ACR) diagnostic criteria
* Subjects who used more than 1 Disease Modifying Antirheumatic Drug (DMARD) including MTX (methotrexate) for 6 months or longer
* Subjects with ESR (erythrocyte sedimentation rate) ≥ 28mm/h or CRP (C-reactive protein)≥ 1.0 mg/dL
* Subjects with ≥ 3 swollen joints out of 66 joints assessed
* Subjects with ≥ 6 tender joints out of 68 joints assessed

Exclusion Criteria:

* Pregnant or nursing women, or subjects who plan to become pregnant within 6 months or whose screening test results show pregnancy cannot be ruled out
* Subjects with previous experience of tacrolimus (excluding external preparations)
* Subjects with renal dysfunction or with serum creatinin > 1.4 mg/dL at screening
* Following subjects with hepatic dysfunction: viral infection, non-viral infection, hepatic cirrhosis, and Serum Glutamic Oxaloacetic Transaminase / Serum Glutamic Pyruvic Transaminase (SGOT/SGPT) exceeding twice the upper limit of normal at screening
* Subjects with pancreatitis, uncontrolled diabetes or complication(s) or with HbA1c > 6.4% at screening
* Subjects complicated with hyperkalemia or with serum potassium level >5.5 mEq/L at screening
* Subjects with history of heart disease (ischemic heart disease, arrhythmia requiring treatment, and heart failure), etc or complications
* Subjects complicated with severe respiratory disease and infection
* Subjects with history of malignant tumor or complication(s) (However, the subjects who are considered to have no risk of recurrence with malignant tumor untreated for 5 years or longer can enter the study. The subjects who succeeded in treatment for basal cell or squamous cell carcinoma of skin can also enter the study.)
* Subjects who were treated with other investigational product(s) within 3 months before screening
* Other subjects who are considered ineligible for the study by the investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2015-05-11 (Actual)

PRIMARY OUTCOMES:
ACR20 response rate 6 months post dose | Baseline and 6 months post dose
  ACR20 is 20% improvement in ACR (American College of Rheumatology) core set

SECONDARY OUTCOMES:
ACR50 response rates at month 6 | Baseline and at month 6
  ACR50 is 50% improvement in ACR (American College of Rheumatology) core set
ACR70 response rates at month 6 | Baseline and at month 6
  ACR70 is 70% improvement in ACR (American College of Rheumatology) core set
Change in DAS28 from baseline to 6 months | Baseline and at month 6
  DAS (Disease Activity Score in Rheumatoid Arthritis)
Change in bone loss rate from baseline to 6 months | Baseline and at month 6
  comparative factors for bone loss rate: bone mineral densitometry [BMD], bone turnover marker test
Safety assessed by the incidence of adverse events, vital signs and lab-tests | For 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- South Korea (4):
  - Busan
  - Daejeon
  - Gyeonggi-do
  - Seoul

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=151